CLINICAL TRIAL: NCT06052046
Title: How Does Total30 for Astigmatism Perform During a Long Day of Wear?
Brief Title: Total30 for Astigmatism Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern College of Optometry (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-00006733
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2023-11

CONDITIONS: Contact Lens Complication; Astigmatism; Refractive Errors
Keywords: TOTAL30 for Astigmatism; Comfort; Dryness; Visual Analog Scale; Contact Lens
MeSH Terms: conditions — Astigmatism; Refractive Errors

STUDY DESIGN:
Intervention Model Description: This prospective, one-month, three-visit study will refit all participants into TOTAL30 for Astigmatism Contact Lenses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Total30 for Astigmatism Contact Lenses (Experimental): TOTAL30 for Astigmatism Monthly Replacement Contact Lenses
  Interventions: Device: TOTAL30 for Astigmatism Contact Lenses

INTERVENTIONS:
Device: TOTAL30 for Astigmatism Contact Lenses — Participants will be refit into TOTAL30 for Astigmatism Contact Lenses and followed for 1 month.
  Other Names: Lehfilcon A

SUMMARY:
Determine if Total30 for Astigmatism contact lenses (CLs) provide a comfortable wearing experience all day. CL discomfort affects most CL wearers with discomfort consistently topping the reasons why established CL wearers drop out of CLs. In fact, studies have consistently found that the frequency of CL dropout is around 20% with this dropout frequency staying relatively stable over the past 20 plus years. This static frequency of CL dropout is surprising since there have been a number of dramatic soft CL innovations during this time frame (e.g., widely available daily disposable CLs, silicone hydrogel CL materials with high oxygen transmissibility, new CL surface coatings).

DETAILED DESCRIPTION:
A common issues that contact lens (CL) wearers frequently face is that their discomfort symptoms increase towards the end of the wear day. This burdensome discomfort can unfortunately cause patients to remove their CLs before their desired wear time. While comfortable wear times vary from patient to patient, Terry et al. has suggested that patients should be able to comfortably wear their CLs for at least 12 hours per day for at least 6 days per week. Nevertheless, the literature currently lacks sufficient data to comment fully on the full day wear experience, which for many patients may be 16 or more hours per day, especially if they have demanding careers. One CL that has the potential to allow for all day comfort is the Total30 for Astigmatism CLs, which is a new water gradient, monthly CL aimed at delivering all day comfort and visual performance. Thus, the purpose of this study is to map comfort over the full wear day in established, asymptomatic, soft CL wearers who are refit in Total30 for Astigmatism CLs. These data are not only important for judging the performance of Total30 for Astigmatism CLs, but they will provide some of the first insights into the full day CL wearing experience over one month.

ELIGIBILITY:
Inclusion Criteria:

* 18- to 45-year-old
* Visual acuity 20/20 or better
* Contact Lens Dry Eye Questionnaire [CLDEQ]-8 scores <10
* Willing to wear Total30 for Astigmatism CLs
* Have a smart phone with text messaging capabilities
* Astigmatism ranging from 0.75 D to 2.50 D in each eye
* Regularly worn 2 week or monthly CLs within the past 6 months
* Current CL wearer
* Glasses prescription that is less than 2 years old
* Willing to start wearing their CLs between 6:00 AM and 8:00 AM and wear their CLs until 11:00 PM each day text messaging data is collected

Exclusion Criteria:

* Current or past hard CL wearers
* A known systemic health condition that is thought to alter tear film physiology
* A history of viral eye disease
* A history of ocular surgery
* A history of severe ocular trauma
* Have an active ocular infection or inflammation
* Currently using isotretinoin-derivatives or ocular medications
* Currently using rewetting drops or artificial tears
* Pregnant or breast feeding
* Willing to discontinue usage of current toric CLs one week prior to the initial visit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Comfort Scores | Change from baseline at 1 month
  A VAS will be used to compare end of day ocular comfort at about 16 hours of contact lens wear (± 50 scale with +50 being best possible comfort and -50 being worst possible comfort).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kannarr Eye Care, Pittsburg, Kansas
  - Coldwater VIsion Center, Coldwater, Mississippi

IPD SHARING:
Plan to Share IPD: No
Summary data will be published in a peer-reviewed manuscript.

REFERENCES:
- [Derived] Lievens C, Perkins A, Rayborn E, Wang Y, Franklin Q, May K, Kannarr S, Bromley M, Pucker AD. Real-Time Changes in the Comfort of a Toric, Monthly, Soft Contact Lens Over a Long Day of Wear. Clin Optom (Auckl). 2024 Dec 17;16:317-325. doi: 10.2147/OPTO.S490934. eCollection 2024. PMID 39713278